CLINICAL TRIAL: NCT05848232
Title: A Prospective Single-Arm Multicenter Study Evaluating Use of the CORA Catheters for the Crossing of Coronary Chronic Total Occlusions
Brief Title: Single-Arm Study Evaluating Use of the CORA Catheters for the Crossing of Coronary Chronic Total Occlusions
Acronym: Cora CTO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ReFlow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-009
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-11

CONDITIONS: Coronary Occlusion
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- coraFlex, coraForce, and/or coraCross Catheters (Experimental): Single arm
  Interventions: Device: coraFlex Catheter; Device: coraForce Catheter; Device: coraCross Catheter

INTERVENTIONS:
Device: coraFlex Catheter — The coraFlex catheter is intended to facilitate the intraluminal placement of conventional guidewires beyond occluded coronary lesions.
Device: coraForce Catheter — The coraForce catheter is intended to facilitate the intraluminal placement of conventional guidewires beyond occluded coronary lesions.
Device: coraCross Catheter — The coraCross catheter is intended to facilitate the intraluminal placement of conventional guidewires beyond occluded coronary lesions.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of the coraFlex, coraForce, and coraCross catheters for crossing chronic total occlusions of the coronary arteries. The study will compare the rate of procedure success to success rates from previous trials.

Participants will undergo percutaneous coronary intervention (PCI) for a chronic total occlusion and be followed for 30 days post-procedure.

DETAILED DESCRIPTION:
The primary objective of this prospective, multicenter, single arm clinical study is to compare the rate of procedure success of the coraCross, coraForce, and coraFlex catheters in facilitating guidewire placement beyond coronary chronic total occlusions to a pre-defined performance goal based on literature. The study population will consist of those 18 years or older with symptomatic ischemic heart disease, undergoing clinically indicated percutaneous recanalization of an occlusive coronary lesion, and meeting all other eligibility criteria. Measures will be assessed through 30 days post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pre-Procedure Inclusion Criteria:

  1. Subject willing and able to provide informed consent and able to comply with the study protocol and follow up.
  2. Male or non-pregnant female ≥18 years of age at time of consent.
  3. Subjects experiencing clinical symptoms suggestive of ischemic heart disease or has evidence of myocardial ischemia attributed to the CTO target vessel and is scheduled for clinically indicated percutaneous revascularization.
  4. Subject is a candidate for PTCA, stenting, and emergency CABG.
* Angiographic Inclusion Criteria:

  1. A minimum of one de novo lesion with at least one target segment in a native coronary vessel meeting CTO criteria {defined as TIMI grade 0 flow} and estimated to be > 3 months duration by clinical history and/or comparison with a prior angiogram or electrocardiogram.

Exclusion Criteria:

* Pre-procedure Exclusion Criteria:

  1. Subject unwilling or unable to comply with the protocol or follow-up requirements, in the opinion of the investigator.
  2. Subject life expectancy less than one year, in the opinion of the investigator.
  3. Subject is pregnant or planning to become pregnant during the course of the trial.
  4. Evidence of MI within 72 hours prior to the index procedure.
  5. History of stroke or transient ischemic attack within 6 months prior to the index procedure.
  6. Prior coronary interventional procedure (including coronary artery bypass graft surgery) of any kind within 30 days of the index procedure.
  7. Inability to tolerate DAPT with aspirin plus a P2Y12 inhibitor.
  8. Known allergies or sensitivities to heparin, antiplatelet drugs, or other anticoagulant therapies, which could not be substituted, including history of major bleeding event in the last 6 months.
  9. Allergy or sensitivity to contrast media that cannot be adequately pre-treated prior to the index procedure.
  10. Subjects with known history of clinically significant abnormal laboratory findings ≤30 days prior to enrollment including:

      1. Neutropenia (<1000 neutrophils/mm3)
      2. Thrombocytopenia (<100,000 platelets/mm3)
      3. AST, ALT, ALP, or bilirubin > 1.5 times ULN
      4. Serum creatinine > 2.0 mg/dL
  11. Subject has signs/symptoms of systemic infection/sepsis (temperature ≥ 38.00 Celsius and WBC ≥12,000 cells/µL). If subject has localized infection or infection is adequately treated and controlled, per investigator discretion, patient may be enrolled.
  12. Evidence of current clinical instability including:

      1. Sustained systolic blood pressure <100 mmHg or cardiogenic shock
      2. Acute pulmonary edema or severe congestive heart failure (NYHA class IV)
      3. Known or suspected acute myocarditis, pericarditis, endocarditis, or cardiac tamponade
      4. Known or suspected dissecting aortic aneurysm
      5. Hemodynamically significant valvular heart disease, hypertrophic cardiomyopathy, restrictive cardiomyopathy, or congenital heart disease.
      6. Requires mechanical circulatory support (e.g., Impella) during index procedure
  13. Subject is currently enrolled in another investigational device or drug trial that interferes with the study endpoints.
  14. Any concurrent, medical, psychological, or social condition which may significantly interfere with the subject's optimal participation in the study, in the opinion of the investigator.
* Angiographic Exclusion Criteria:

  1. Target lesion is located within a stent (in-stent occlusion).
  2. Target vessel has other lesions proximal to the total occlusion with >75% stenosis (based on visual estimate) unless there is planned stenting of the proximal lesion as well.
  3. Angiography demonstrates extensive lesion related thrombus (TIMI thrombus grade 3 or 4).
  4. Fractured stents in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Procedure success defined as technical success and the absence of in-hospital Major Adverse Cardiovascular Events (MACE) | Through hospital discharge or 24 hours post-procedure (whichever comes first)
  * Technical success is defined as angiographic confirmation of chronic total occlusion crossing with guidewire placement, facilitated by one or more of the Cora Catheters, in the target vessel true lumen either distal or proximal to the occlusion, depending on the route of access.
  * MACE includes cardiac death, myocardial infarction {Q-wave or non-Q-wave, with CK-MB >3 times upper limit of normal}, and target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Azzalini, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No